CLINICAL TRIAL: NCT04443621
Title: Changes in the Perception of Personal Dignity Over the Course of Dementia
Acronym: DIDEM
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Palacky University (Other)
Collaborators: University Hospital Hradec Kralove (Other); Faculty Hospital Kralovske Vinohrady (Other Government); University Hospital Olomouc (Other); University Hospital Ostrava (Other)
Responsible Party: Principal Investigator, Helena Kisvetrova, Principal Investigator, Palacky University
Other Study IDs: NU20-07-00100
Record Dates: First submitted 2020-06-19; First posted 2020-06-23 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Dementia; Dignity
Keywords: dignity; dementia; older adult; perception
MeSH Terms: conditions — Dementia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- participants with early stage dementia: Subjects with diagnosed any type of dementia at an early phase (MMSE score 20 - 25 points) - for longitudinal study (three phasis).
  Interventions: Behavioral: questionnaire; Behavioral: in-depth interview
- participants without dementia: Subjects without dementia with MMSE score 26 - 30 points (for validation of ACE-III).
  Interventions: Behavioral: questionnaire

INTERVENTIONS:
Behavioral: questionnaire — Questionnaire battery for assessment of dignity, cognition, self-sufficiency, and depression.
Behavioral: in-depth interview — Individual in-depth interviews with OAwD on the topic of dignity (two interviews with each respondent at a 12-month interval) .
  Groups: participants with early stage dementia

SUMMARY:
Dignity is an integral part of quality of life (QoL). Older adults often face with situations that are related with the development of dementia and that might significantly affect their feeling of personal dignity. The aim of the project is to investigate the changes in the perception of personal dignity amongst older adults with dementia (OAwD) over the course of three years and to define factors that threaten their dignity. A mixed methods design (longitudinal prospective study) will be used. In the quantitative part, a battery of Czech questionnaires will be used, and a translation and validation of a Czech version of the ACE-III will be carried out. The qualitative part will include in-depth interviews (narrative and semi-structured). The sample will comprise of OAwD living in home setting. Knowledge of the changes in the perception of personal dignity and related factors may aid the healthcare staff in choosing interventions that support and preserve dignity of OAwD as a significant part of their QoL. The project is a follow-up of a previous project No. 16-28628A.

DETAILED DESCRIPTION:
A. Introduction to project, current state of art As the population ages, an increasing number of people will be diagnosed with dementia. At present, there are some 47 million people living with dementia worldwide. In Czech Republic, there are about 156,000 people suffering from dementia. Regional estimates of dementia prevalence in people aged 60 years and over now range from 4.6% in Central Europe to 8.7% in North Africa and the Middle East. It is estimated up to 131 million people with dementia will live in the world by 2050. Thus, there is a need of sensitive and specific cognitive assessment tools to detect cognitive impairment. It enables to provide timely intervention to delay the disease progression, prolong independence, and enhance the quality of life (QoL) and personal dignity of the individual with dementia.

Dementia is neurodegenerative disease characterized by progressive, irreversible and still incurable cognitive decline. People suffering from dementia retain their positive personality traits and character. However, as the illness progresses, symptoms such as memory loss, speech impairment, disorientation, difficulties with activities of daily living, and self-neglect are common. This leads to a significant interference with everyday social and work activities and has a negative impact on subjective perception of dignity. At present, the Mini Mental State Examination (MMSE) is used in the Czech Republic to diagnose dementia. Due to copyright issues with the MMSE (similar to the Montreal Cognitive Assessment [MoCA] questionnaire), there is a need for another valid tool to be free available in the country. Currently, the most frequently used tool in the world is the Addenbrooke's Cognitive Examination III (ACE-III), which is composed of five domains: orientation and attention; memory; fluency; language, and visuospatial function. The ACE-III-J is a sensitive and specific screening test to diagnose dementia, and it was better than the MMSE in accuracy for identifying dementia.

Dignity is described as an integral part of QoL. Similarly to QoL, dignity can also be understood as a multidimensional concept including: dignity of identity (self-worth/worthiness, integrity, trust); dignity as a human right (equality, freedom of choice); and dignity as expression of autonomy (independence, control. There are three main dimensions essential for constituting dignity: A historical dignity-dimension, acknowledging one's own life projects and history; an intrapersonal dignity-dimension, recognizing one's own human worth, and living according to individual values; and an interpersonal dignity-dimension, experiencing being part of a caring and confirming society.

Jacobson (2007) says that dignity exists in two complementary, yet disparate forms. It is understood as a dualistic concept incorporating absolute and relative dignity, objective and subjective dignity, and personal and social dignity. Personal dignity is a type of dignity that is subjectively perceived by an individual and is linked to a sense of worthiness. However, personal dignity is also contingent and contextual, and can be influenced both by an internal aspect, which is the worth and self-respect one ascribes to oneself, as well as by an external aspect, which is the worth and value ascribed to the individual by others.

Patients with a severe chronic disease (such as neurodegenerative) experience existential concerns related to changes in the self because of the disease, as well as the social consequences of the disease (e.g. embarrassment, role changes, loss of independence, and stigmatization), which can severely affect the sense of personal dignity.

Older adults with dementia (OAwD) are often experiencing an ongoing loss of personal dignity, value and security, and experiencing cognitive decline can be a threat towards self-respect and the sense of dignity. The key element of the dementia experience is the effort to preserve one's identity or sense of self and to preserve a meaningful life. Multiple personal losses and changes such as increased dependency, loss of autonomy and gradual loss of abilities or competencies can have a negative impact on the sense of self and the self-esteem of dementia sufferers. Thus, OAwD are in risk of personal dignity loss due to both impact of the disease on their identity and self-esteem, and indirectly through negative social interactions and experiences. Before entering the stage of severe dementia individuals are aware of the progressive decline in their abilities and actively try to cope with this decline. A sound sense of personal dignity is essential to the individual's overall experience of well-being and his/her QoL. Investigation of the factors that maintain and strengthen personal dignity needs to incorporate data collected from those afflicted. However, research how having dementia may impact personal dignity into person's subjective experience of mild to moderate dementia is only very recent.

Pilot data The proposed grant project builds on results of a previous project Trajectories of quality of life by the elderly in in early-stage dementia (No. 16-28628A). The findings of the project confirm that OAwD assess their QoL better when they have a greater sense of personal dignity. The validated Czech version of Patient Dignity Inventory (PDI-CZ) created and tested in our project No. 16-28628A will be used in the proposed project.

B. Project objectives, project timeline and description of methods and approaches To define the factors that pose a threat to personal dignity gives an opportunity for a deeper understanding of these issues. This can subsequently assist healthcare staff with choosing the optimum interventions supporting QoL amongst OAwD. The proposed project responds to a society-wide need to identify and solve psychosocial needs of an ageing population with emphasis on neurodegenerative diseases.

The objective of the project is to investigate the changes in the perception of personal dignity of OAwD. The opportunity to define risk factors threatening personal dignity over the course of dementia will contribute to a deeper understanding of patients' needs. This will help healthcare workers choose the optimum psychosocial interventions in accordance with Evidence Based Practice and thus protect dignity of OAwD as a major component of QoL. This may have a positive effect on the psycho-social dimension of QoL amongst OAwD and may lower the frequency and length of hospitalizations as well as save costs on healthcare and social services.

The main aim is to ascertain how the subjective perception of personal dignity in OAwD changes throughout the course of this disease (trajectory of personal dignity perception) and which factors affect it. Because different types of dementia might have different perceptions of personal dignity related to specific disturbances of cognitive domains, post-hoc subgroup analysis in different forms of dementia will be performed. For the assessment of cognition and diagnosis of dementia, the Addenbrooke's Cognitive Examination III (ACE-III), POBAV, and ALBA questionnaires will be used. For this reason, we need to create and validate a Czech version of the ACE-III as the first stage of the project.

In order to achieve the main aim, five sub-aims were identified which should make it possible to ascertain subjective perception of personal dignity and factors which affect in amongst OAwD:

1. to create a Czech version of the ACE-III and to conduct a psychometric validation;
2. to ascertain how the assessment of personal dignity changes over the course of 2 years;
3. to identify sociodemographic and clinical factors perceived as a threat to dignity;
4. post-hoc subgroup analysis of results among the different types of dementia;
5. to define the differences in the perception of personal dignity among OAwD when using quantitative (PDI-CZ) and qualitative (in-depth interview) methods.

C. Methodology In order to reach the set aims, a mixed methods research design (quantitative survey first follow by qualitative interview) will be used to carry out a longitudinal, prospective study.

In the quantitative phase of the project using a battery of standardized questionnaires (3 stages). Research nurse gave QAwD the questionnaires and explained how to complete them. The questionnaires will be completed on project enrolment and then two more times at a 12-month interval.

In the qualitative phase of the research, individual in-depth interviews with OAwD on the topic of dignity (two interviews with each respondent at a 12-month interval) will be conducted, recorded, and transcribed with a subsequent interpretative phenomenological analysis. Two psychologists will be undertaking the interviews, in order to ensure that the interviews are conducted in the most sensitive manner. Informed consent will be secured before each interview. This will be carried out throughout project lifetime.

Questionnaire battery will be included: Addenbrooke's Cognitive Examination III (ACE-III), Amnesia Light and Brief Assessment (ALBA), POBAV, Patient Dignity Inventory (PDI-CZ), Bristol Activities of Daily Living Scale (BADLS-CZ), Geriatric Depression Scale (GDS), and a batch of socio-demographic and clinical characteristics (including age, sex, level of education, living arrangement, social life, frequency of social visits, telephone contact with relatives/friends, and the daytime spent alone, illnesses, medication, etc).

Sample The sample will consist of community-dwelling (i.e., living at home) older adults. They will be addressed together with their family caregivers in neurologic and geriatric outpatient offices.

Sample size:

First sample (quantitative research) will comprise of 500 respondents (310 OAwD for the longitudinal, three-stage study and 190 older adults for the validation study ACE-III).

Second sample (qualitative research) - after evaluating the 1st stage of the quantitative research, we will select 10 OAwD from the sample group with high level (average scale more than 3) and 10 OAwD who have low level of dignity to understand the different perspectives of perception of personal dignity. The exact number of respondents will depend on the thematic saturation in the course of interviewing.

Data from the quantitative research (validation study, and longitudinal study) will be gathered using a questionnaire from 310 OAwD (longitudinal study) and 190 older adults (half with dementia and half without dementia; validation study ACE-III) in neurologic and geriatric outpatients' departments in four regions of the Czech Republic. All data will be inserted into CASTOR database, from which they will be exported for statistical processing.

Data from the qualitative phase will be gathered using in-depth interviews with 20 OAwD. These respondents we will select after evaluation the 1st stage of the quantitative research (10 OAwD with high and 10 OAwD with low levels of dignity to understand the different perspectives in perception of personal dignity). An interpretative phenomenological analysis (IPA) will be applied. The IPA is an approach of a qualitative research, which is used to examine how people make sense of their major life experiences. The method is often used to study patients' lived experience. The data will be coded in NVivo 12 software for analysis. To assure reliability of the analysis, two researchers will code the interviews independently and they will confront their results for similarities and differences.

ELIGIBILITY:
Inclusion Criteria:

* Group I.: age ≥60 years; lives at home; diagnosed with dementia (MMSE score 20 - 25 points), ability to consent to participate in the research; in contact with a family caregiver at least once a week.
* Group II: age ≥60 years; lives at home; MMSE score 26 - 30 points, ability to consent to participate in the research.

Exclusion Criteria:

* for both groups: severe psychotic disorder; severe cognitive impairment (severe hearing, visual or speech impairment), and terminal stage of caner or non-cancer disease.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Older adults aged ≥60 years.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Addenbrooke's Cognitive Examination III (ACE-III) | 12 months
  To create a Czech version of the ACE-III and to conduct a psychometric validation
Patient Dignity Inventory (PDI) | 24 months
  To ascertain how the assessment of personal dignity changes over the course of two years
Factors affecting dignity | 24 months
  To identify sociodemographic and clinical factors perceived as a threat to dignity (including age, sex, level of education, living arrangement, social life, frequency of social visits, telephone contact with relatives/friends, and the daytime spent alone, illnesses, depression, self-sufficiency etc).
Differences in the perception of personal dignity | 24 months
  To define the differences in the perception of personal dignity among OAwD when using quantitative (PDI-CZ) and qualitative (in-depth interview) methods.

SECONDARY OUTCOMES:
Dignity among the different types of dementia | 24 months
  Post-hoc subgroup analysis of results among the different types of dementia

CONTACTS AND LOCATIONS:
Overall Officials: Helena Kisvetrova, PhD, Principal Investigator — Faculty of Health Sciences Palacky University Olomouc
Locations (5):
- Czechia (5):
  - University Hospital Hradec Kralove, Hradec Králové
  - Palacky University, Olomouc
  - University Hospital Olomouc, Olomouc
  - University Hospital Ostrava, Ostrava
  - Faculty Hospital Kralovske Vinohrady, Prague

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kisvetrova H, Bretsnajdrova M, Juraskova B, Langova K. Personal dignity in people with early-stage dementia: A longitudinal study. Nurs Ethics. 2024 Nov;31(7):1258-1270. doi: 10.1177/09697330241244495. Epub 2024 Apr 5. PMID 38578289
- [Derived] Kluzova Kracmarova L, Tomanova J, Cernikova KA, Tavel P, Langova K, Greaves PJ, Kisvetrova H. Perception of dignity in older men and women in the early stages of dementia: a cross-sectional study. BMC Geriatr. 2022 Aug 18;22(1):684. doi: 10.1186/s12877-022-03362-3. PMID 35982424